CLINICAL TRIAL: NCT06662383
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of Retatrutide Compared to Tirzepatide in Adults Who Have Obesity
Brief Title: A Study of Retatrutide (LY3437943) Compared to Tirzepatide (LY3298176) in Adults Who Have Obesity
Acronym: TRIUMPH-5
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18585; J1I-MC-GZBP (Other: Eli Lilly and Company); 2024-511450-49-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — retatrutide; Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Retatrutide (Experimental): Participants will receive retatrutide administered subcutaneously (SC)
  Interventions: Drug: Retatrutide
- Tirzepatide (Active Comparator): Participants will receive tirzepatide administered SC
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Retatrutide — Administered SC
  Other Names: LY3437943
  Arms: Retatrutide
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of retatrutide compared to tirzepatide in adults who have obesity. The study will last about 89 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have obesity and a history of at least one self-reported unsuccessful dietary effort to reduce body weight.

Exclusion Criteria:

* Have a self-reported change in body weight >5 kilograms (kg) (11 pounds) within 90 days before screening.
* Have a prior or planned surgical treatment for obesity.
* Have a prior or planned endoscopic procedure and/or device-based therapy for obesity.
* Have taken weight loss drugs, including over-the-counter medications, within 90 days prior to screening.
* Have a family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2).
* Have had within the past 90 days before screening:

  * acute myocardial infarction
  * cerebrovascular accident (stroke)
  * coronary revascularization
  * hospitalization for unstable angina, or
  * hospitalization due to congestive heart failure.
* Have New York Heart Association Functional Classification Class IV congestive heart failure.
* Have a history of chronic or acute pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 80

SECONDARY OUTCOMES:
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 80
Change from Baseline in Waist Circumference | Baseline, Week 80
Percent Change from Baseline in Total Cholesterol | Baseline, Week 80
Percent Change from Baseline in Triglycerides | Baseline, Week 80
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 80
Change from Baseline in Diastolic Blood Pressure (DBP) | Baseline, Week 80
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 80
Percent Change from Baseline in Fasting Insulin | Baseline, Week 80
Change from Baseline in Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) | Baseline, Week 80

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (65):
- United States (40):
  - Medical Advancement Centers of Arizona, Tempe, Arizona
  - Mary & Dick Allen Diabetes Center, Newport Beach, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Lynn Institute of Denver, Aurora, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Encore Medical Research, Hollywood, Florida
  - Suncoast Research Group, Miami, Florida
  - Onhealth Research Center, Miami, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Einstein Clinical Research, Vero Beach, Florida
  - ClinCept Clinical Research - MH, Columbus, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Pivotal Research Solutions, Stonecrest, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Great Lakes Research Institute, Southfield, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Las Vegas Endocrinology, Henderson, Nevada
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - New York Gastroenterology Associates, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - PharmQuest Life Sciences, LLC, Greensboro, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - PriMED Clinical Research, Dayton, Ohio
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - Headlands Horizons LLC, Brownsville, Texas
  - Next Level Urgent Care, Houston, Texas
  - Houston Research Institute, Houston, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
- Argentina (5):
  - DIM Clínica Privada, Ramos Mejía, Buenos Aires
  - Centro Médico Viamonte, Buenos Aires, Buenos Aires F.D.
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires, Buenos Aires F.D.
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires, Buenos Aires F.D.
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
- Germany (9):
  - Gemeinschaftspraxis Prof. Dr. med. Stephan Jacob, Dr. med. Frohmut Jacob, Villingen-Schwenningen, Baden-Wurttemberg
  - Diabetologische Schwerpunktpraxis Dr. Staudenmeyer & Dr. Schiwietz, Lingen, Lower Saxony
  - Zentrum fur klinische Forschung - Köln, Cologne, North Rhine-Westphalia
  - InnoDiab Forschung Gmbh, Essen, North Rhine-Westphalia
  - Medizentrum Essen Borbeck, Essen, North Rhine-Westphalia
  - AmBeNet GmbH, Leipzig, Saxony
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Diabetes Zentrum Wilhelmsburg, Hamburg
  - Diabeteszentrum Hamburg West, Hamburg
- Poland (10):
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan, Greater Poland Voivodeship
  - Nzoz Neuro-Kard Ilkowski i Partnerzy SPL, Poznan, Greater Poland Voivodeship
  - Gabinety TERPA, Lublin, Lublin Voivodeship
  - Ekamed, Lublin, Lublin Voivodeship
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok, Podlaskie Voivodeship
  - Gabinet Leczenia Otylosci i Chorob Dietozaleznych - dr hab. n. med. Lucyna Ostrowska, Bialystok, Podlaskie Voivodeship
  - Zdrowie Osteo-Medic, Bialystok, Podlaskie Voivodeship
  - NZOZ Specjalistyczny Ośrodek Internistyczno-Diabetologiczny, Bialystok, Podlaskie Voivodeship
  - NZOZ Przychodnia Specjalistyczna Andrzej Wittek, Henryk Rudzki, Ruda Śląska, Silesian Voivodeship
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz, Łódź Voivodeship
- Ponce Medical School Foundation Inc., Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Retatrutide (LY3437943) Compared to Tirzepatide (LY3298176) in Adults Who Have Obesity (TRIUMPH-5) — https://trials.lilly.com/en-US/trial/549215